CLINICAL TRIAL: NCT02099682
Title: Takepron Capsules 15/ Orally Dispersing (OD) Tablets 15 Special Drug Use Surveillance Long-term Use Survey on the Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Low-dose Aspirin
Brief Title: Long-term Use of Takepron Capsules on the Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Low-dose Aspirin
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 467-712; JapicCTI-142414 (Registry Identifier: JapicCTI); JapicCTI-R150735 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Gastric or Duodenal Ulcers
Keywords: Pharmacological therapy
MeSH Terms: conditions — Duodenal Ulcer | interventions — Lansoprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lansoprazole 15 mg: Lansoprazole 15 mg orally once daily
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole Capsules 15/ OD Tablets
  Other Names: Takepron Capsules 15/ OD Tablets

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of long-term administration of lansoprazole (Takepron) for up to 12 months in the routine clinical setting in patients receiving low-dose aspirin

DETAILED DESCRIPTION:
This is a special survey on long-term use (for up to 12 months) of lansoprazole (Takepron) to determine the incidence of adverse drug reactions in the routine clinical setting in patients receiving low-dose aspirin.

The usual adult dosage is 15 mg of lansoprazole administered orally once daily.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with a history of gastric or duodenal ulcers (2) Patients requiring long-term use of low-dose aspirin (81-324 mg once daily) as prophylaxis for thromboembolism (3) Patients taking low-dose oral aspirin (81-324 mg once daily) at the start of administration of lansoprazole (including patients who start low-dose aspirin on the same day as the start of administration of lansoprazole)

Exclusion Criteria:

* (1) Patients with gastric or duodenal ulcer (in the active [A1, A2] or healing [H1, H2] stage if assessed endoscopically) at the start of administration of lansoprazole (2) Patients with active upper gastrointestinal hemorrhage at the start of administration of lansoprazole (3) Patients with contraindications for lansoprazole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastric or duodenal ulcers
Sampling Method: Non-Probability Sample
Enrollment: 3366 (Actual)
Dates: Start 2010-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 460 investigative sites in Japan from August 2010 to January 2014 (N=3366).
Pre-assignment Details: Patients with a history of gastric or duodenal ulcers and requiring long-term use of low-dose aspirin were enrolled in the study.
Period: Overall Study
Arm/Group | Lansoprazole 15 mg
Started | 3366 (Number of cases.)
Safety Analysis Set (SAS) | 3255 (All participants who took the study drug at least once.)
Completed | 3255
Not Completed | 111
Not completed — Data Not Available | 51
Not completed — Lost to Follow-up | 31
Not completed — Other | 29

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all participants who took the study drug at least once.
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3255
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1399
  Male | 1856
Purpose for Low-Dose Aspirin Use [Number; unit: participants] — Participants could be counted in more than 1 category.
  participants
    Angina pectoris | 1182
    Myocardial infarction | 531
    Transient ischaemic attack (TIA) | 221
    Cerebral infarction | 1225
    Post-coronary artery bypass (CABG) | 106
    PTCA | 398
    Other | 316
Gastric or Duodenal Ulcer History Breakdown [Number; unit: participants] — Participants could be counted in more than 1 category.
  participants
    Gastric ulcer | 2718
    Duodenal ulcer | 313
    Unknown | 252
Gastric or Duodenal Ulcer History: Time of Onset [Number; unit: participants]
  Within 6 months of study drug administration | 213
  ≥ 6 months, < 1 year before start of treatment | 138
  1 year or longer before the start of treatment | 977
  Unknown | 1927
H. pylori infection [Number; unit: participants]
  Negative | 425
  Positive | 171
  Unknown | 2659

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Drug Reactions
Description: Frequency, severity, and time to onset of adverse drug reactions tabulated by each symptom. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: 12 months
Population: Safety analysis set - All participants who received at least 1 dose of lansoprazole.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3255
participants
  Enteritis infectious | 1
  Lymphoma | 1
  Diabetes mellitus | 1
  Anxiety | 1
  Dizziness | 2
  Dysgeusia | 1
  Headache | 1
  Loss of consciousness | 1
  Sudden hearing loss | 1
  Abdominal discomfort | 1
  Abdominal distension | 1
  Abdominal pain | 1
  Colitis | 1
  Constipation | 2
  Diarrhoea | 23
  Enterocolitis | 1
  Gastrooesophageal reflux disease | 1
  Haematochezia | 1
  Nausea | 4
  Colitis microscopic | 3
  Hypoaesthesia oral | 1
  Faeces soft | 1
  Drug eruption | 3
  Eczema | 1
  Hypersensitivity vasculitis | 1
  Pruritus | 1
  Rash generalised | 1
  Back pain | 1
  Osteoporosis | 1
  Renal failure chronic | 1
  Sudden death | 1
  Thirst | 1
  Hepatic enzyme increased | 1
  Glycosylated haemoglobin increased | 1
  Weight decreased | 1
  Fall | 1
  Spinal fracture | 1

2. Secondary Outcome: Presence or Absence of Endoscopic Examinations
Description: Summary of data on the presence or absence of endoscopic examinations.
Time Frame: From baseline to 12 months
Population: Efficacy analysis set: all participants who took the study drug at least once excluding those with gastric ulcers or duodenal ulcers at initiation of study drug treatment, or participants for whom low-dose aspirin use during study drug treatment could not be confirmed.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  With endoscopy | 2773
  Without endoscopy | 437

3. Secondary Outcome: Presence of Gastric or Duodenal Ulcer
Description: Summary of data on the presence or absence of gastric or duodenal ulcers.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  Present | 3190
  Absent | 20

4. Secondary Outcome: Presence of Gastric or Duodenal Hemorrhagic Lesion
Description: Summary of data on the presence or absence of gastric or duodenal hemorrhagic lesions.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  Present | 3201
  Absent | 9

5. Secondary Outcome: Presence of Either Gastric/Duodenal Ulcer, or Gastric/Duodenal Hemorrhagic Lesion
Description: Summary of data on the presence or absence of gastric/duodenal ulcer gastric/duodenal hemorrhagic lesion.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  Present | 3186
  Absent | 24

6. Secondary Outcome: Treatment for Gastric/Duodenal Ulcer or Lesion
Description: Summary of data on the presence or absence of treatment for duodenal ulcers or hemorrhagic lesions.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  Present | 0
  Absent | 24

7. Secondary Outcome: Details of Treatment (Including Duplicates) for Gastric or Duodenal Ulcers or Hemorrhagic Lesions
Description: Summary of data on the details of treatment for gastric or duodenal ulcers or hemorrhagic lesions.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  Takepron Capsule or OD Tablet 15 mg | 15
  Takepron Capsule or OD Tablet 30 mg | 2
  Rabeprazole tablet 10 mg | 2
  H2 receptor antagonist (oral) | 1
  Omeprazole (injection) | 2
  H2 receptor antagonist (injection) | 1
  Other peptic ulcer drugs | 2
  Endoscopic hemostasis | 1
  Other | 5

8. Secondary Outcome: Treatment Outcome (Including Duplicates) for Gastric or Duodenal Ulcers or Hemorrhagic Lesions
Description: Summary of data on the outcome of treatment for gastric or duodenal ulcers or hemorrhagic lesions.
Time Frame: From baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg
Number analyzed (Participants) | 3210
participants
  Takepron 15 mg: Recovery | 9
  Takepron 15 mg: Relief | 6
  Takepron 30 mg: Recovery | 1
  Takepron 30 mg: Relief | 1
  Rabeprazole 10 mg: Recovery | 1
  Rabeprazole 10 mg: Relief | 1
  H2 receptor antagonist (orally): Recovery | 1
  H2 receptor antagonist (orally): Relief | 1
  Omeprazole (injection): Recovery | 1
  Omeprazole (injection): Relief | 1
  H2 receptor antagonist (injection): Recovery | 2
  H2 receptor antagonist (injection): Relief | 1
  Other peptic ulcer drugs: Recovery | 3
  Other peptic ulcer drugs: Relief | 2
  Endoscopic hemostasis: Recovery | 9
  Endoscopic hemostasis: Relief | 6
  Other: Recovery | 1
  Other: Relief | 1

ADVERSE EVENTS:
Time Frame: From the first dose of open-label study drug until 14 days (or 30 days for a serious adverse event) after the last dose of open-label study drug (up to 12 months).
Description: Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Arm/Group | Lansoprazole 15 mg
Serious Adverse Events (participants affected / at risk) | 126/3225
Other Adverse Events (participants affected / at risk) | 0/3255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole 15 mg (N=3225)
Appendicitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pyelonephritis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Agitation (Psychiatric disorders) | 1
Psychosomatic disease (Psychiatric disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 5
Convulsion (Nervous system disorders) | 1
Dyslalia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Angina pectoris (Cardiac disorders) | 4
Angina unstable (Cardiac disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 8
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 6
Myocardial infarction (Cardiac disorders) | 5
Ventricular arrhythmia (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 3
Aortic dissection (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Aortic rupture (Vascular disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Gastric polyps (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileal ulcer (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Death (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Accidental device ingestion (General disorders) | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Coronary angioplasty (Surgical and medical procedures) | 1
Enterostomy (Surgical and medical procedures) | 1
Cardiac failure chronic (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.